CLINICAL TRIAL: NCT03310437
Title: Cost Effectiveness of Primary PCI Versus Thrombolytic Therapy in STEMI in Assiut University Hospital
Brief Title: Cost Effectiveness if Primary PCI Versus Thrombolytic Therapy in Acute STEMI in Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nahed Sameh Zaki (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Nahed Sameh Zaki, Principle investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 81
Record Dates: First submitted 2017-09-25; First posted 2017-10-16 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary PCI: In primary PCI we use arterial sheath , wires ,heparin ,intracoronary stents
  Interventions: Procedure: Primary PCI
- Thrombolytic: In patients recieving thrombolytics they continue on LWMH for 72h ,plus aspirin , clopedogril , BB, statins

INTERVENTIONS:
Procedure: Primary PCI — Primary percutaneous coronary intervention in acute myocardial infarction patients
  Groups: Primary PCI

SUMMARY:
Cost effectiveness between PPCI and thrombolytic therapy in STEMI patients without contraindications

DETAILED DESCRIPTION:
Cost effectiveness between PPCI and thrombolytic therapy in STEMI patients 100 patient each within 90 m for PPCI and 6h for thrombolytic

ELIGIBILITY:
Inclusion Criteria:

* All PPCI patients within 90 minutes door to ballon.
* All thrombolytic patient without contraindication ,within 6 golden hours of chest pain.

Exclusion Criteria:

* patients don't meet inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presented by ST elevation myocardial infarction
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Compare between PPCI and thrombolytic therapy regarding over all cost in STEMI patients | one year for collecting 100 patient for each arm with follow up 6 month
  we will compare different outcomes in ST elevation myocardial infarction patients presented to our hospital who had recieved intervention (primary PCI ) versus thrombolytic as regarded in all over cost in egyptian pounds and follow up for 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut medicine faculty, Asyut, Egypt